CLINICAL TRIAL: NCT05434689
Title: Phase Ib/II Trial Of Iberdomide-Combinations In Patients With Positive Minimal Residual Disease (>10-5) After Autologous Hematopoietic Cell Transplantation In The Upfront Management Of Patients With Multiple Myeloma
Brief Title: COMbination Regimens in MM Post AHCT to elimiNate MRD Utilizing IbERdomide
Acronym: COMMANDER
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bristol-Myers Squibb (Industry); coMMit Myeloma Trials (Unknown)
Responsible Party: Principal Investigator, Luciano Jose Costa, MD, Professor of Medicine, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB-21113; Amgen, Inc (Other: Amgen, Inc.); BMS (Other: BMS)
Record Dates: First submitted 2022-06-10; First posted 2022-06-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; daratumumab; Dexamethasone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Iberdomide, Daratumumab and Dexamethasone (Regimen A) (Experimental): Iberdomide dosed according to cohort assignment days 1-21. Dexamethasone 40 mg oral or intravenously (20 mg for participants 70 or older) on days 1,8,15 and 22 Darartumumab and hyalurnonidase-fihj 1,800mg/30,000 units subcutaneously on days 1,8,15,22 (cycles 1,2) or on days 1,15 (cycles 3-6)
  Interventions: Drug: Iberdomide; Drug: Daratumumab; Drug: Dexamethasone
- Iberdomide, Carfilzomib, Daratumumab and Dexamethasone (Regimen B) (Experimental): Iberdomide dosed according to cohort assignment days 1-21. Dexamethasone 40 mg oral or intravenously (20 mg for participants 70 or older) on days 1,8,15 and 22 Darartumumab and hyalurnonidase-fihj 1,800mg/30,000 units subcutaneously on days 1,8,15,22 (cycles 1,2) or on days 1,15 (cycles 3-6) Carfilzomib dosed intravenously dosed according to cohort assignment on days 1, 8, 15 (Consistent with standard practice, the very first dose of carfilzomib (cycle 1 day 1) must be 20 mg/m^2).
  Interventions: Drug: Iberdomide; Drug: Daratumumab; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Iberdomide — Iberdomide (Iber, CC-220) is a novel cereblon E3 ligase modulator (CELMoD) in development for treatment of multiple myeloma and other conditions.
Drug: Daratumumab — Anti-CD 38 monoclonal antibody established in the treatment of multiple myeloma
Drug: Dexamethasone — Corticosteroid active against multiple myeloma in combination with other agents
Drug: Carfilzomib — Second generation proteasome inhibitor with activity in multiple myeloma
  Arms: Iberdomide, Carfilzomib, Daratumumab and Dexamethasone (Regimen B)

SUMMARY:
Similar to the paradigm established in other hematologic malignancies that are considered curable, the achievement of MRD(-) status is necessary for long term disease control in MM. The fact that the majority of patients remain MRD (+) after induction therapy and AHCT points to the opportunity to deploy novel agents with complementary mechanism of action and favorable toxicity profile to reach and maintain MRD (-) status.

Given its favorable toxicity profile, the convenience of oral administration, and compelling single agent activity even in heavily pretreated MM, iberdomide is likely amenable to long term therapy in patients with high-risk of relapse/progression identified by the persistence of MRD(+). The investigators intend to develop combination(s) of iberdomide with other agents with complementary mechanism of action in the consolidation setting post AHCT in order to achieve and sustain MRD (-).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years with no upper age limit
2. Confirmation of newly diagnosed multiple myeloma (MM) with 1-2 prior regimens utilized in induction that included an immunomodulatory agent (IMiD) and a proteasome inhibitor (PI) combined or in different regimens
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
4. Prior AHCT 100-180 days prior to initiation of protocol-directed therapy
5. MRD ≥ 10^-5 by clonoSEQ® NGS platform, determined 60-120 days after AHCT as part of the usual care.
6. No prior disease progression (either before or since AHCT)
7. Overall response (i.e post-AHCT compared to historical baseline prior to initiation of any therapy for MM) ≥ PR.
8. Measurable disease at the time of the initial diagnosis (i.e. prior to starting any therapy for MM) meeting at least one of the following criteria:

   * Serum monoclonal (M) protein ≥1.0 g/dl

     * 200 mg of M protein/24h in the urine
   * Difference between involved and uninvolved free light chain ≥10 mg/dL and abnormal kappa to lambda ratio.
9. Adequate hepatic function evidenced by AST and ALT ≤ 3 x ULN and bilirubin ≤ 1.5 ULN.
10. Adequate bone marrow function evidenced by platelets ≥ 75,000 /mm3 (without transfusion of platelets in the prior 7 days) and absolute neutrophil count ≥ 1,000/mm3.
11. Creatinine clearance (CrCl) ≥ 40 mL/minute within 28 days prior to start of therapy either measured or calculated using standard Cockcroft and Gault formula (available in https://www.kidney.org/professionals/KDOQI/gfr_calculatorCoc ).
12. Females of childbearing potential (FCBP) must have two negative pregnancy tests as verified by the investigator and agree to ongoing pregnancy testing and to practice contraception during treatment. Male subjects must agree to practice contraception and refrain from donating sperm during treatment.
13. In line with the higher incidence of MM in Blacks, and to address the historical underrepresentation of ethnical minorities in MM trials, at least 25% of the enrolled patients will be of ethnical minorities.
14. Written informed consent in accordance with federal, local, and institutional guidelines.

Exclusion Criteria:

1. Diagnosis of amyloidosis, POEMS, Waldenstrom's macroglobulinemia, plasma cell leukemia or smoldering multiple myeloma (i.e. never evolved to active myeloma).
2. Major surgery or radiotherapy within 28 days of starting protocol-directed treatment.
3. Acute active infection requiring treatment within 14 days of starting protocol-directed treatment.
4. Current or prior involvement of central nervous system by multiple myeloma.
5. MM refractory to prior CD38 monoclonal antibody therapy and/or to carfilzomib (prior exposure allowed). Refractoriness here is defined as not achieving at least a PR in a regimen containing the agent or disease progression < 60 days from last dose of the agent.
6. Pregnant or lactating females.
7. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
8. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
9. Unstable angina or myocardial infarction within 4 months prior to starting protocol-directed treatment, NYHA Class II, III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker.
10. A prolongation of QT interval on screening electrocardiogram (ECG) as defined by corrected QT interval (QTc) > 480 ms using Fridericia's QT correction formula.
11. Cerebrovascular disease manifested as prior stroke at any time or TIA in the 12 months prior to initiation of therapy.
12. Uncontrolled hypertension (per investigator assessment, despite optimal medical management)
13. Diagnosis of interstitial lung disease
14. Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or localized thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas.
15. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 28 days prior to starting protocol-directed treatment.
16. For regimen B - Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
17. Contra indication or intolerance to required supportive care medications (Aspirin and Acyclovir)
18. Concomitant use of strong inhibitors or inducers of CYP3A4, P-gp, or BCRP, or BCRP substrate with a narrow therapeutic index, for at least 14 days or 5 half-lives (whichever is shorter). (consult https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers )
19. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent Diagnosis of amyloidosis, POEMS, Waldenstrom's macroglobulinemia.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | One year
  Proportion of patients in each regimen who develop dose limiting toxicity
MRD conversion ( to < 10-5 MM-associated molecules) | Four years
  Rate MRD conversion ( to <10-5 MM-associated molecules) at completion of consolidation therapy. Patients who are not assessed for MRD at the completion of consolidation (due to any reason, including death, withdrawal from study, loss to follow-up, missed assessment, etc) will be considered as not having achieved MRD conversion.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Costa, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Duke University, Durham, North Carolina
  - Ohio State University Medical College, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt University Medical College, Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided